CLINICAL TRIAL: NCT04203264
Title: Real-Time Identification of Gastric Lesions and Anatomical Landmarks During Magnetically Controlled Capsule Endoscopy Using Artificial Intelligence
Brief Title: Real-Time Identification System of Magnetically Controlled Capsule Endoscopy Using Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Other Study IDs: 20190411A
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Capsule Endoscopy
Keywords: artificial intelligence; magnetically controlled capsule endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Real-time artificial intelligence identification system — The patients swallowed the MCE with a small amount of water in the left lateral decubitus position. Once the capsule reached the stomach after investigating the esophagus, it was lifted away from the posterior wall, rotated and advanced to the fundus and cardiac regions, and then to the gastric body, angulus, antrum and pylorus. The magnetic steering time for passing through the pylorus was not allowed more than 15 min. The real-time auxiliary system implemented real-time processing for the output image of MCE system. Professional operators guarantee the integrity of the examination and the diagnostic results of professional endoscopist was used as the gold standard. The system diagnosis results was recorded at the same time. The sensitivity, delay time, specificity of lesions and anatomical landmarks will be analyzed.

SUMMARY:
The aim of this study is to evaluate the performance of real-time auxiliary system based on artificial intelligence algorithm in lesion detection and quality control in magnetically controlled capsule endoscopy.

DETAILED DESCRIPTION:
Magnetically controlled capsule endoscopy (MCE) has been used in clinical practice for gastric examination, with high sensitivity and specificity of 90.4% and 94.7%, respectively.

Therefore, a real-time auxiliary system based on convolutional neural network deep learning framework was developed to assist clinicians to improve the quality in MCE examinations.

Patients referred for magnetically controlled capsule endoscopy (MCE) in the participating center were prospectively enrolled. After passage through the esophagus, physician will finish the gastric examination under magnetic steering with the real-time auxiliary system. Professional operators guarantee the integrity of the examination and the diagnostic results of professional endoscopist was used as the gold standard. The system diagnosis results was recorded at the same time. The sensitivity, delay time, specificity of lesions and anatomical landmarks will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* With or without gastrointestinal complaints
* Scheduled to undergo a capsule endoscopy for both stomach and small bowel
* Signed the informed consents before joining this study

Exclusion Criteria:

* Dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy
* Refused abdominal surgery to take out the capsule in case of capsule retention
* Implanted pacemaker, except the pacemaker is compatible with MRI
* Other implanted electromedical devices or magnetic metal foreign bodies
* Pregnancy or suspected pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients undergoing magnetically controlled capsule endoscopy examination
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-16 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | up to 2 weeks
  The sensitivity of lesions detected by system

SECONDARY OUTCOMES:
Delay time | up to 2 weeks
  Average preprocessing and displaying times before and after the execution of system
Specificity | up to 2 weeks
  The specificity of detected by system
Accuracy of anatomic landmarks identification | up to 2 weeks
  Accuracy of anatomic landmarks ( cardia, fundus, body, lesser curvature, greater curvature, angle, antrum and pylorus) identified by real-time identification system
Completeness of real-time observation with assistance | up to 2 weeks
  Whether the clinician observed all anatomic landmarks of stomach (cardia, fundus, body, angulus, antrum and pylorus).
Accuracy of heat map | up to 2 weeks
  The rate of the highlighted area indicated in the lesion
Lesion detection yield | up to 2 weeks
  The ratio of lesions detected by system to all lesions

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Wu L, Zhang J, Zhou W, An P, Shen L, Liu J, Jiang X, Huang X, Mu G, Wan X, Lv X, Gao J, Cui N, Hu S, Chen Y, Hu X, Li J, Chen D, Gong D, He X, Ding Q, Zhu X, Li S, Wei X, Li X, Wang X, Zhou J, Zhang M, Yu HG. Randomised controlled trial of WISENSE, a real-time quality improving system for monitoring blind spots during esophagogastroduodenoscopy. Gut. 2019 Dec;68(12):2161-2169. doi: 10.1136/gutjnl-2018-317366. Epub 2019 Mar 11. PMID 30858305
- [Background] Ding Z, Shi H, Zhang H, Meng L, Fan M, Han C, Zhang K, Ming F, Xie X, Liu H, Liu J, Lin R, Hou X. Gastroenterologist-Level Identification of Small-Bowel Diseases and Normal Variants by Capsule Endoscopy Using a Deep-Learning Model. Gastroenterology. 2019 Oct;157(4):1044-1054.e5. doi: 10.1053/j.gastro.2019.06.025. Epub 2019 Jun 25. PMID 31251929